CLINICAL TRIAL: NCT05398146
Title: The Effect of Listening to Music, Performing Mathematics Operations and Ball Squeezing in Reducing Pain During Dressing Change in Children With Appendectomy
Brief Title: The Effect of Three Methods Used in Reducing Pain During Dressing Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Yilmaz Akdag (Other)
Collaborators: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Melike Yilmaz Akdag, Principal Investigator, RN, MSc, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018.5.07
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: pain; appendectomy; child; distraction; dressing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Dressing (Experimental): Information about the children and their parents who agreed to participate in the study was recorded on the 'Information Form' 5 minutes before the dressing procedure by the researcher.
  Interventions: Behavioral: mathematical operations; Behavioral: ball squeezing; Behavioral: listening to music; Other: kontrol grubu
- During Dressing (Experimental): The first dressing of all children included in the study after appendectomy was performed by the doctor in the clinic. No distraction method was applied to the children in the control group during dressing. The children in the LM group were dressed while listening to music. The children in the BS group continued to squeeze the ball during the dressing. The children in the MO group were asked to perform mathematical operations given by the nurse. While the dressing was in progress, the pulse and oxygen saturation levels were recorded in the information form by the nurse. At the last stage of dressing, the children were asked to mark the level of pain they experienced during dressing on the VAS, immediately after the sticking plaster was placed on the surgical area. Parents and nurses assessed the pain level of the child during dressing through the VAS.
  Interventions: Behavioral: mathematical operations; Behavioral: ball squeezing; Behavioral: listening to music; Other: kontrol grubu
- Post-Dressing (Experimental): When the dressing was over, the application of distraction methods was terminated. After the dressing, the child's pulse and oxygen saturation levels were recorded in the information form by the nurse.
  Interventions: Behavioral: mathematical operations; Behavioral: ball squeezing; Behavioral: listening to music; Other: kontrol grubu

INTERVENTIONS:
Behavioral: mathematical operations — Prepared by the researchers, the form involved mathematical operations such as addition, subtraction, multiplication, and division. The difficulty level of the mathematical operations in the form was determined by age groups of children. Accordingly, mathematical operations were divided into 3 groups primary school, secondary school and high school levels.
Behavioral: ball squeezing — For the children in the BS group, a softball that could fit in the palm and be easily squeezed by the child was used.
Behavioral: listening to music — Children were allowed to listen to music with headphones during dressing changes.
Other: kontrol grubu — No application was made during dressing change in children. Routine dressing change of the clinic was applied.

SUMMARY:
This randomized controlled study aims to determine the effect of listening to music (LM), ball squeezing (BS), and performing mathematical operations (MO) in reducing the pain experienced during the first dressing in children aged 8-18 with appendectomy.

DETAILED DESCRIPTION:
The sample of the study consisted of 120 children (LM:30, BS:30, MO:30, control:30). A minute before dressing and during dressing, the children in the LM group listened to music, the children in the SB group squeezed the ball, the children in the MO group performed mathematical operations.According to the child, parent, and nurse assessment, it was determined that the mean pain score of the children in the LM and MO groups was lower than that of the BS group and control groups (p< .05).

ELIGIBILITY:
Inclusion Criteria:

* Consisted of the child and parent's consent to participate in the study,
* The child and parent's speaking Turkish at the level of native speaker,
* The child's being 8-18 years old and undergoing appendectomy,
* Being the body temperature of the child in the normal level (36.5-37.2⁰C),
* The child's not having intense nausea and vomiting,
* The child's not having any physical, intellectual or neurological disability that would affect his/her participation.

Exclusion Criteria:

* Having a mental or neurological disability
* Children with hearing and vision impairment

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Pain Scores pre-dressing | 60 seconds
  Visual Analog Scale (VAS) was used for determine pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
Comparison of Pain Scores During Dressing | 60 seconds
  Visual Analog Scale (VAS) was used for determine pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
Comparison of Pain Scores post-Dressing | 60 seconds
  Visual Analog Scale (VAS) was used for determine pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).

CONTACTS AND LOCATIONS:
Overall Officials: birsen mutlu, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No